CLINICAL TRIAL: NCT06685835
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Efficacy and Safety of Brensocatib in Adults With Moderate to Severe Hidradenitis Suppurativa - The CEDAR Study
Brief Title: A Study of the Efficacy and Safety of Brensocatib in Adults With Moderate to Severe Hidradenitis Suppurativa (HS)
Acronym: CEDAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1007-231; 2024-515959-38-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: HS
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Brensocatib 10 mg (Experimental): Participants will receive brensocatib 10 mg tablet, once daily (QD), orally for 52 weeks.
  Interventions: Drug: Brensocatib
- Brensocatib 40 mg (Experimental): Participants will receive brensocatib 40 mg tablet, QD, orally for 52 weeks.
  Interventions: Drug: Brensocatib
- Placebo Followed by Brensocatib 10 mg (Placebo Comparator): Participants will receive brensocatib-matching placebo tablet, QD, orally for 16 weeks, and then Brensocatib 10 mg tablet, QD, orally for 36 weeks.
  Interventions: Drug: Brensocatib; Drug: Placebo
- Placebo Followed by Brensocatib 40 mg (Placebo Comparator): Participants will receive brensocatib-matching placebo tablet, QD, orally for 16 weeks, and then Brensocatib 40 mg tablet, QD, orally for 36 weeks.
  Interventions: Drug: Brensocatib; Drug: Placebo

INTERVENTIONS:
Drug: Brensocatib — Film-coated Oral tablet
  Other Names: INS1007
Drug: Placebo — Film-coated Oral tablet
  Arms: Placebo Followed by Brensocatib 10 mg; Placebo Followed by Brensocatib 40 mg

SUMMARY:
The primary purpose of the study is to evaluate the effect of brensocatib compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS (confirmed by a dermatologist), with a history of signs and symptoms consistent with HS for at least 6 months before the Screening Visit.
* Moderate or severe HS defined as a total of ≥6 inflammatory lesions (inflammatory nodules and/or abscesses) for at least 8 weeks before the Baseline Visit.
* HS lesions in at least 2 distinct anatomic areas, 1 of which must be at least Hurley Stage II or Hurley Stage III at both the Screening and Baseline Visits.

Exclusion Criteria:

* Draining tunnel count of ≥20 at the Baseline Visit.
* Surgical or laser intervention for an HS lesion during the Screening Period.
* Clinical diagnosis of Papillon-Lefèvre Syndrome.
* Participants with an absolute neutrophil count <1,000/mm3 at the Screening Visit.
* Participants having active liver disease or hepatic dysfunction.
* Have diagnosed periodontal disease under active management by a dentist or expected to have periodontal disease-related procedures within the study period.
* Received systemic (intravenous or orally [PO]) antibiotic therapy within 8 weeks before the Baseline Visit

  a. Doxycycline or minocycline up to 100 mg twice daily is permitted provided the dosing regimen being stable for at least 8 weeks before the Baseline Visit and is expected to continue.
* Received PO or transdermal opioid analgesics (except tramadol) for any reason within 4 weeks before the Baseline Visit.
* Permitted analgesics for HS-related pain have not been at a stable dose regimen for at least 4 weeks before the Baseline Visit.
* Received prescription topical therapies for the treatment of HS within 2 weeks before the Baseline Visit.
* Received any anti-tumor necrosis factor (TNF)-α/other biologics treatment within 12 weeks or 5 elimination half-lives, whichever is longer, before the Baseline Visit.
* Received systemic nonbiologic therapies (eg, corticosteroids and retinoids) for HS within 4 weeks before the Baseline Visit.
* Received any immunomodulatory agents within 4 weeks before the Baseline Visit.

Note: Other Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2027-01-28 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Total Abscess and Inflammatory Nodule (AN) Count at Week 16 | Baseline and Week 16

SECONDARY OUTCOMES:
Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) at Week 16 | Week 16
Percentage of Participants Achieving HiSCR75 at Week 16 | Week 16
Percentage of Participants Achieving ≥2-point Decrease From Baseline in Hidradenitis Suppurativa - Investigator's Global Assessment (HS-IGA) at Week 16 | Week 16
Change From Baseline in Draining Tunnel Count at Week 16 | Baseline and Week 16
Percentage of Participants Remaining Free from HS Flare by Week 16 | Week 16
Change From Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) Score at Week 16 | Baseline and Week 16
Percentage of Participants Achieving IHS4-55 at Week 16 | Week 16
Change From Baseline on Dermatology Life Quality Index (DLQI) Global Score at Week 16 | Baseline and Week 16
Percentage of Participants Achieving Numeric Rating Scale 30 (NRS30) at Week 16 with a Baseline NRS Score ≥3 | Week 16
Number of Participants who Experienced at Least One Adverse Event (AE) | Up to Week 56
Plasma Concentration of Brensocatib | Pre-dose and at multiple timepoints post-dose up to Week 56

CONTACTS AND LOCATIONS:
Locations (72):
- United States (26):
  - USA001, Phoenix, Arizona
  - USA007, Sacramento, California
  - USA026, Coral Gables, Florida
  - USA027, Hollywood, Florida
  - USA021, Margate, Florida
  - USA018, Miami, Florida
  - USA025, Ocala, Florida
  - USA004, Tampa, Florida
  - USA010, Weston, Florida
  - USA028, Atlanta, Georgia
  - USA011, Sandy Springs, Georgia
  - USA003, Plainfield, Indiana
  - USA002, Baton Rouge, Louisiana
  - USA017, Boston, Massachusetts
  - USA012, Detroit, Michigan
  - USA024, Fort Gratiot, Michigan
  - USA020, Minneapolis, Minnesota
  - USA015, St Louis, Missouri
  - USA013, Lebanon, New Hampshire
  - USA009, Cleveland, Ohio
  - USA016, Springfield, Ohio
  - USA019, Hershey, Pennsylvania
  - USA022, Philadelphia, Pennsylvania
  - USA005, Dallas, Texas
  - USA023, Dallas, Texas
  - USA008, Spokane, Washington
- Australia (5):
  - AUS003, Darlinghurst, New South Wales
  - AUS004, Kogarah, New South Wales
  - AUS001, Brisbane, Queensland
  - AUS006, Woolloongabba, Queensland
  - AUS002, Fremantle, Western Australia
- Bulgaria (4):
  - BGR001, Lovech
  - BGR003, Pleven
  - BGR004, Sofia
  - BGR002, Stara Zagora
- Canada (7):
  - CAN003, Barrie, Ontario
  - CAN006, Guelph, Ontario
  - CAN007, Peterborough, Ontario
  - CAN011, Richmond Hill, Ontario
  - CAN009, Richmond Hill, Ontario
  - CAN010, Toronto, Ontario
  - CAN004, Québec
- France (5):
  - FRA001, Lyon, Auvergne-Rhône-Alpes
  - FRA004, Toulouse, Haute-Garonne
  - FRA002, Antony
  - FRA003, Paris
  - FRA005, Rouen
- Germany (6):
  - DEU007, Langenau, Baden-Wurttemberg
  - DEU002, Darmstadt, Hesse
  - DEU001, Bochum, North Rhine-Westphalia
  - DEU003, Dresden, Saxony
  - DEU006, Dessau-RoÃŸlau
  - DEU005, Lübeck
- Greece (4):
  - GRC002, Athens, Attica
  - GRC004, Chaïdári, Attica
  - GRC001, N. Efkapria-Pavlos Melas, Thessaloniki
  - GRC003, Thessaloniki
- NLD001, Rotterdam, Netherlands
- Poland (8):
  - POL006, Wroclaw, Lower Silesian Voivodeship
  - POL008, Warsaw, Masovian Voivodeship
  - POL002, Rzeszów, Podkarpackie Voivodeship
  - POL004, Krakow
  - POL007, Warsaw
  - POL001, Warsaw
  - POL005, Wroclaw
  - POL003, Wroclaw
- Spain (6):
  - ESP006, Badalona, Barcelona
  - ESP004, Las Palmas de Gran Canaria, Las Palmas Provincia
  - ESP001, Manises, Valencia
  - ESP002, Madrid
  - ESP005, Madrid
  - ESP003, Madrid

IPD SHARING:
Plan to Share IPD: No